CLINICAL TRIAL: NCT05770674
Title: Prospective, Open-label, Multicenter, Randomized Clinical Trial Comparing 1 Month vs. 12 Months Dual Antiplatelet Therapy in Patients Undergoing Percutaneous Coronary Intervention With Genoss® Drug Eluting Stent
Brief Title: Comparison of 1 Month vs. 12 Months DAPT in Patients Undergoing PCI With Genoss® DES
Acronym: GENOSS-DAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kiyuk Chang (Other)
Collaborators: Uijeongbu St. Mary Hospital (Other); St Vincent's Hospital (Other); Bucheon St. Mary's Hospital (Other); Wonju Severance Christian Hospital (Other); Chungbuk National University Hospital (Other); Daejeon St. Mary's hospital (Other); Korea University Guro Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Kiyuk Chang, MD, PhD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC21MIDI0023
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Dual Antiplatelet Therapy; Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Month DAPT (Active Comparator): Patients will receive 300 mg of aspirin and 300 mg of clopidogrel before PCI unless previously medicated with antiplatelet agents. Aspirin 100 mg plus clopidogrel 75 mg once daily will be given for 1 month following PCI. Following 1 month, clopidogrel 75 mg once daily will be given for 11 months.
  Interventions: Drug: 1 Month vs. 12 Months DAPT
- 12 Months DAPT (Active Comparator): Patients will receive 300 mg of aspirin and 300 mg of clopidogrel before PCI unless previously medicated with antiplatelet agents. Aspirin 100 mg plus clopidogrel 75 mg once daily will be given for 12 months following PCI.
  Interventions: Drug: 1 Month vs. 12 Months DAPT

INTERVENTIONS:
Drug: 1 Month vs. 12 Months DAPT — Dual antiplatelet therapy with aspirin plus clopidogrel will be given for the following period after PCI according to patient allocation
  1. 1 Month following PCI, followed by clopidogrel monotherapy
  2. 12 Months following PCI

SUMMARY:
This study is a prospective, open-label, multicenter, randomized clinical trial to evaluate the efficacy of 1 month dual antiplatelet therapy (DAPT) with aspirin plus clopidogrel followed by clopidogrel monotherapy, compared with 12 months DAPT with aspirin plus clopidogrel in patients undergoing percutaneous coronary intervention with Genoss® drug eluting stents.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 inhibitor is recommended following percutaneous coronary intervention (PCI). However, the optimal duration of DAPT is still controversial, and current US and European guidelines recommend 12+ months for Acute Coronary Syndrome (ACS) and 6+ months in Chronic Coronary Syndrome (CCS). A meta-analysis comparing short (6 months) and long-term (12 months) DAPT has shown a lower risk of bleeding with no significant increase in ischemia risk associated with short DAPT use.

Monotherapy with a P2Y12 inhibitor clopidogrel has been proposed as a novel alternative to DAPT in patients with atherosclerotic cardiovascular disease. Clopidogrel has shown comparable bleeding events after PCI compared to aspirin, and reduced the risk of subsequent ischemic events. In addition, several trials have reported that clopidogrel monotherapy now has a lower risk of bleeding than antiplatelet drug therapy (DAPT). These results suggest that P2Y12 inhibitor monotherapy has a lower risk of bleeding in patients with PCI and can be compared with DAPT in preventing recurrent ischemic events.

Given that Genoss® Drug-Eluting Stent (DES) has a very low incidence of Stent Thrombosis (ST), short-term DAPT after PCI is now expected to reduce the risk of bleeding with clopidogrel instead of aspirin, without increasing cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 19 years of age
* Subjects undergoing elective PCI with Genoss® Drug Eluting Stents
* Subject who can understand the risk, benefit and treatment alternatives, and when he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure

Exclusion Criteria:

* Subjects presenting with acute myocardial infarction
* Subjects with less than 1 year of life expectancy
* Subjects presenting with cardiogenic shock
* Subjects requiring anticoagulation (warfarin, direct oral anticoagulant), or those requiring antiplatelet agents other than aspirin and P2Y12 inhibitors.
* Subjects with history of intracranial hemorrhage (ICH)
* Known hypersensitivity or contraindications to study medications (aspirin, clopidogrel), or drugs used in the procedure (heparin, contrast media, sirolimus). Those with contrast hypersensitivity can be enrolled if symptom/signs can be controlled by anti-histamines or steroids.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2186 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NACE (Net Adverse Clinical Event) | 12 Months
  A composite of cardiovascular death, myocardial infarction, ischemic or hemorrhagic stroke, definite stent thrombosis, or BARC (Bleeding Academic Research Consortium) type 3 or 5 bleeding events

SECONDARY OUTCOMES:
MACE (Major Adverse Cardiovascular Events) | 12 Months
  A composite of cardiovascular death, myocardial infarction, ischemic or hemorrhagic stroke, or definite stent thrombosis
BARC Type 3 / 5 bleeding events | 12 Months
  Bleeding defined by BARC types 3 or 5
All cause death | 12 Months
  Death by any cause
Cardiovascular death | 12 Months
  Death by cardiac cause
Myocardial infarction | 12 Months
  Myocardial infarction
Ischemic or hemorrhagic stroke | 12 Months
  Ischemic or hemorrhagic stroke
Definite or probable stent thrombosis | 12 Months
  Definite or probable stent thrombosis
Any revascularization | 12 Months
  Any repeat revascularization
Ischemia-driven target lesion revascularization | 12 Months
  Ischemia-driven repeat revascularization of target lesion
BARC Type 2/3/4/5 bleeding | 12 Months
  Bleeding defined by BARC types 2, 3, 4, or 5
BARC Type 3/4/5 bleeding | 12 Months
  Bleeding defined by BARC types 3, 4, or 5

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea